CLINICAL TRIAL: NCT03005223
Title: Drug-Drug Interaction Study Between DWC20155 / DWC20156 and DWC20163 in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DW_DWJ1366005
Record Dates: First submitted 2016-12-26; First posted 2016-12-29 (Estimated); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Healthy

ARMS (2):
- Study effect of DWC20163 on DWC20155/DWC20156 PK (Experimental): To study effect of DWC20163 on DWC20155/DWC20156 PK
  Interventions: Drug: Co-administration of DWC20155/DWC20156; Drug: DWC20163
- Study effect of DWC20155/DWC20156 on DWC20163 PK (Experimental): To study effect of DWC20155/DWC20156 on DWC20163 PK
  Interventions: Drug: Co-administration of DWC20155/DWC20156; Drug: DWC20163

INTERVENTIONS:
Drug: Co-administration of DWC20155/DWC20156
Drug: DWC20163

SUMMARY:
A randomized, open label, crossover study to explore drug-drug interactions between DWC20155 / DWC20156 and DWC20163 in Healthy Volunteers

ELIGIBILITY:
Inclusion Criteria:

* Accepts healthy volunteers

Exclusion Criteria:

* Who has allergy to investigational product

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2017-01-04 (Actual); Primary Completion 2017-05 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | 0 ~ 24 hours
Area under the time versus plasma concentration curve (AUC) | 0 ~ 24 hours